CLINICAL TRIAL: NCT01324544
Title: A Multicenter, Inpatient, Open-label Study to Characterize the Pharmacokinetics, Safety, and Efficacy of Intravenous Dosing of Buprenorphine in Pediatric Patients Aged From Birth to 6 Years of Age (Inclusive) Who Require Opioid Analgesia for Acute Moderate to Severe Pain
Brief Title: Pharmacokinetics, Safety, and Efficacy of Intravenous Dosing of Buprenorphine in Pediatric Patients Who Require Opioid Analgesia for Acute Moderate to Severe Pain
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to change in development plan.
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUP3030; 2010-021955-14 (EudraCT Number)
Record Dates: First submitted 2011-03-24; First posted 2011-03-29 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Other Acute Postoperative Pain; Prolonged Endotracheal Intubation
Keywords: Acute Pain; Opioid; Analgesia
MeSH Terms: conditions — Acute Pain; Agnosia | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Buprenorphine IV (Experimental): Buprenorphine IV
  Interventions: Drug: Buprenorphine IV

INTERVENTIONS:
Drug: Buprenorphine IV — Buprenorphine IV administered via patient-controlled analgesia (PCA) pump for at least 24 hours and up to 72 hours.
  Other Names: Buprenex

SUMMARY:
The purpose of this study is to characterize the safety, pharmacokinetics (PK), and efficacy of intravenous (IV) buprenorphine in pediatric patients.

DETAILED DESCRIPTION:
A study of the PK, safety, and efficacy of IV buprenorphine in acute moderate to severe pain in male and female pediatric patients aged from birth to 6 years, inclusive, requiring continuous opioid analgesic treatment for at least 24 hours and up to 72 hours.

ELIGIBILITY:
Inclusion Criteria include:

* Must have written informed consent provided by the parent or legal guardian and/or patient assent, when appropriate
* Male and female children, from birth to aged 6 years, inclusive, with minimum weight of 2.5 kg
* Have or are anticipated to have acute moderate to severe pain; requiring treatment with an intravenous (IV) opioid analgesic medication for at least 24 hours postoperatively or; due to prolonged endotracheal intubation requiring IV opioid analgesic treatment for at least 24 hours poststabilization
* Must have stable vital signs
* Must have stable respiratory status
* Must be inpatient for the treatment period of the study

Exclusion Criteria include:

* Have any known allergy or sensitivity to buprenorphine or other opioids (this criterion does not include patients who have experienced common opioid side effects [eg, nausea, constipation])
* Have evidence of impaired renal function
* Have hepatic impairment
* Have history of seizures
* Have a history of sleep apnea within the past year
* Have structural heart disease or a pacemaker
* Have clinically unstable cardiac disease
* Have used any investigational medication/therapy within 30 days prior to the first dose of study drug
* Are deemed to be unsuitable by the investigator for reason(s) not specifically stated in the exclusion criteria.

Other protocol-specific inclusion/exclusion criteria may apply.

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measures are clearance (CL/F) and apparent central volume of distribution (Vc/F) estimated using standard population nonlinear mixed effects methodology. | Up to 24 hours

SECONDARY OUTCOMES:
The number of participants with adverse events as a measure of safety. | Up to 10 days